CLINICAL TRIAL: NCT03528564
Title: A Randomized Double-Blinded Phase II Study to Determine Treatment Protocol for Hemoglobin Optimization to Prevent Transfusion and Adverse Events in Perioperative Patients With Iron Restricted Anemia
Brief Title: Hemoglobin Optimization to Prevent Transfusion and Adverse Events in Perioperative Patients With Iron Restricted Anemia
Acronym: HOPE-Hb
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary reasoning is that we were unable to demonstrate feasibility, prior to and because of the impact of COVID on our research programs.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOPE-Hb
Record Dates: First submitted 2018-04-09; First posted 2018-05-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Anemia, Iron Deficiency; Anemia of Chronic Disease; Hip Arthropathy; Knee Arthropathy
Keywords: Preoperative Anemia; Intravenous Iron; Erythropoietin
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Epoetin alfa (Experimental): Preoperative treatment of anemia with iron sucrose (Venofer) plus Epoetin Alfa (Eprex)
  Interventions: Drug: Iron sucrose; Drug: Epoetin Alfa
- Intravenous Iron (Placebo Comparator): Preoperative treatment of anemia with iron sucrose (Venofer) plus placebo (saline)
  Interventions: Drug: Iron sucrose; Drug: Placebo

INTERVENTIONS:
Drug: Iron sucrose — Intravenous iron to be administered to all patients (9 x 5 mL Single Dose Vials @ 20mg elemental iron/mL; 900 mg total)
  Other Names: Venofer
Drug: Epoetin Alfa — Erythropoietin to be administered to half of study participants (40,000 IU x 1-2 subcutaneous injections)
  Other Names: Eprex
  Arms: Epoetin alfa
Drug: Placebo — Saline to be administered to half of study participants (equal volume to Eprex x 1-2 subcutaneous injections)
  Other Names: Saline
  Arms: Intravenous Iron

SUMMARY:
The HOPE-Hb trial is a phase II study to determine the feasibility and impact of a combination treatment (intravenous iron plus erythropoietin) versus intravenous iron treatment alone on preoperative hemoglobin concentration before hip or knee arthroplasty.

DETAILED DESCRIPTION:
The purpose of the HOPE-Hb trial is to determine the feasibility and efficacy of intravenous iron plus erythropoietin versus intravenous iron alone for the treatment of iron restrictive anemia (iron deficiency anemia and anemia of chronic inflammation) prior to unilateral total hip or knee arthroplasty surgery. Half of the study population will be randomly assigned to receive intravenous iron (Venofer; iron sucrose) and Eprex (subcutaneous epoetin alfa), while the other half will be randomized to receive Venofer (intravenous iron sucrose) and placebo (subcutaneous saline). This trial will be conducted in two phases. The vanguard phase will be conducted at a single site with a primary outcome of evaluating feasibility of the study. The full study phase will be conducted at four sites with a primary outcome of determining the impact of a combination treatment (intravenous iron plus erythropoietin) versus intravenous iron treatment alone on preoperative hemoglobin concentration. This study will also examine the RBC transfusion rate and clinical outcomes such as death, stroke, myocardial infarction, pulmonary embolism, infection, kidney injury, and deep vein thrombosis as secondary outcomes.

Preoperatively, patients will be administered a total of 900mg of intravenous iron (Venofer, iron sucrose) over three visits (3-6 weeks before surgery). Then patients will be randomized to receive either two administrations of 40,000 IU of Erythropoietin (Eprex; Epoeitin alfa) or an identical placebo (saline) over two study visits (2-3 weeks before surgery). Study participants will be followed-up for 12 weeks after surgery.

Study assessments and potential adverse events reporting will be undertaken at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of consent
* Undergoing unilateral total hip or knee arthroplasty surgery (primary)
* Hemoglobin concentration of less than 120g/L; but greater than 60g/L

Exclusion Criteria:

* Anemia attributed to something other than iron deficiency anemo/ACI:
* Any other diagnosed or suspected cause of anemia (e.g. macrocytic anemia , lead toxicity, myelodysplastic syndrome)
* Suspected of having acute blood loss due to any diagnosed condition (e.g. malignancy or gastric ulcer)
* Mean Cell Volume (MCV) > 97fL
* Known deficiency of vitamin B12 and/or folate
* A known history of acquired iron overload, haemochromatosis, thalassemia or other hereditary hemoglobinopathy.
* Received an erythropoiesis stimulating agent, IV iron therapy, or red blood cell transfusion in the previous 12 weeks (from the time of consent), or planned use prior to operation
* Blood pressure measured at >180mmHg systolic or >100mmHg diastolic
* Known current or prior history of liver disease or elevation of alanine transaminase (ALT), or aspartate transaminase (AST) more than two times the upper limit of normal
* A known hypersensitivity to IV iron or erythropoietin alfa (Eprex)
* Renal dialysis (current or historical)
* Active infection (currently receiving antibiotics)
* Not eligible for venous thromboembolism prophylaxis
* Prior history of seizures or medical conditions associated with a predisposition to seizure activity such as central nervous system infections and brain metastases
* History of thromboembolic disease or active coronary artery disease
* Women who are pregnant or lactating (women of childbearing potential must be surgically sterile, or more than 1 year postmenopausal, or else must have a negative pregnancy test prior to randomization)
* Recipient of an investigational drug within the past 30 days
* Inability to speak, read, or understand the English language (required for cognitive testing)
* Participation in a preoperative autologous blood donation program for current operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Vanguard Phase (Initial 12 patients): Feasibility of using Erythropoietin + Intravenous Iron to Treat Preoperative Iron Restrictive Anemia | 18 weeks from randomization
  The primary outcome of the vanguard phase is to determine the feasibility of using erythropoietin + intravenous iron to treat preoperative iron restrictive anemia. Feasibility will be measured according to subject enrollment rates, with adherence to the treatment schedule of >80%.
Full Study: Preoperative Hemoglobin Concentration | 6 weeks from randomization
  The primary outcome of the full study is preoperative hemoglobin concentration, as measured on the day of surgery in patients with iron restricted anemia.

SECONDARY OUTCOMES:
Post-Treatment Hemoglobin Concentration | 12 weeks from randomization
  Change in post-treatment hemoglobin concentration from baseline
Change in Hemoglobin Concentration from Initiation of Treatment | 6 weeks from randomization
  Rate of hemoglobin change from initiation of treatment to final preoperative hemoglobin
Postoperative Hemoglobin Concentration | 0 weeks from surgery and 12 weeks from surgery
  Hemoglobin concentration on postoperative day 2 (prior to hospital discharge); and 4-6 weeks after surgery
Red Blood Cell Transfusions | 6 weeks from surgery
  Rate of RBC transfusion and number of units transfused during surgery and up to 6 weeks postoperatively
Deep Vein Thrombosis | 12 weeks from surgery
  Incidence of DVT up to 12 weeks postoperatively
Composite of Morbidity | 3 months from surgery
  Incidence of a composite clinical outcome including death, stroke, myocardial infarction, pulmonary embolism, infection, acute kidney injury, and deep vein thrombosis from treatment to up to 3 months post surgery
Surgical Wound Infection | 6 weeks from surgery
  Incidence of superficial and deep wound infection from treatment to 4-6 weeks post surgery
Assessment of Iron Status | 6 weeks from surgery
  Hematological outcomes for treatment efficacy including: Hb, ferritin, hepcidin, and transferrin saturation (TSAT) pre-operatively and 4-6 weeks postoperatively
Digit Span Test | 6 weeks from surgery
  Cognitive assessment of memory span
California Verbal Learning Test | 6 weeks from surgery
  Cognitive assessment of word learning, recall and recognition, as well as episodic memory
Neuropsychological Impairment Scale | 6 weeks from surgery
  A subjective cognitive assessment of cognitive functioning. This is a 95-item questionnaire, with all items rated on a scale from 0 (not at all) to 5 (extremely). From the 95 total items, 80 items describe neurophysiological symptoms (Global measure of impairment; GMI), 10 items describe affective disturbance, and 5 items assess test-taking attitudes. A total GMI score can range from 0-320, with higher scores indicating an increased impairment index.
Trail Making Test | 6 weeks from surgery
  Cognitive assessment of processing speed
Digit Symbol | 6 weeks from surgery
  Cognitive assessment of response speed, sustained attention, and visual spatial skills
Montreal Cognitive Assessment | 6 weeks from surgery
  Cognitive assessment of global cognitive functioning
Stroop Colour and Word Test | 6 weeks from surgery
  Cognitive assessment of processing speed
Wisconsin Card Sorting Test | 6 weeks from surgery
  Cognitive assessment of a participant's ability to set-shift (display flexibility in the face of changing conditions)
Hospital Anxiety and Depression Scale | 6 weeks from surgery
  Cognitive assessment of anxiety and depression levels. A total score between 0-7 indicates normal levels of depression or anxiety; a total score between 8-10 indicates borderline abnormal levels of anxiety or depression; and a total score between 11-21 indicates abnormal levels of depression or anxiety
Cost Analysis | 12 weeks from randomization
  Assessment of relative cost of treatment and cost savings associated with transfusion avoidance will be assessed (see projected cost analysis; appended)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory MT Hare, MD PhD, Principal Investigator — St. Michael's Hospital; University of Toronto
Locations (1):
- St. Michael's Hosptial, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided